CLINICAL TRIAL: NCT01306409
Title: Neocytolysis in the Treatment of Renal Anemia With Erythropoieses Stimulating Agents
Brief Title: Neocytolysis in the Treatment of Renal Anemia With Erythropoieses Stimulating Agents (ESA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 362/09
Record Dates: First submitted 2011-02-15; First posted 2011-03-01 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Renal Anemia
Keywords: anemia; kidney disease
MeSH Terms: conditions — Anemia; Kidney Diseases | interventions — continuous erythropoietin receptor activator; Darbepoetin alfa; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Sequential application of different ESA
  Interventions: Drug: cera, darbepoetin, epoetin-beta; Drug: ESA

INTERVENTIONS:
Drug: cera, darbepoetin, epoetin-beta — Epoetin once/ 2wk, cera once/ month, darbepoetin once/ 2wk
Drug: ESA — Sequential application of three different ESA

SUMMARY:
The purpose of this study is to gain information on reticulocyte neocytolysis in patients treated with ESA with regard to different types of ESA.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age > 18 years, dialysis dependent chronic renal failure
* hemodialysis three times a week
* Kt/V > 1,2 od URR > 65%
* hemoglobin between 11 and 13 g/dl within the last 2 months
* hemoglobin change +/- 1g/dl within the last 4 weeks
* ESA for at least 8 weeks
* Ferritin > 300 ng/ml and Tsat > 25%

Exclusion Criteria:

* Significant bleeding in the last 8 weeks
* blood transfusion within the last 8 weeks
* hemoglobin disorder
* hemolysis
* Malignant disease
* Significant inflammation
* Acute infection
* CRP > 30 mg/l
* Temporary vascular dialysis access
* Vitamin B12 deficiency
* Folic acid deficiency
* Not controlled hyperparathyroidism
* Not controlled hypertension
* Epilepsia within thze last 6 months
* Thrombocyte count > 500 x 10^9 /l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Reticulocyte count on day 7 | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickenmann, MD, Principal Investigator — Transplantation immunology and nephrology, unversity hospital Basel, Switzerland
Locations (1):
- Nephrology and Transplantaton Immunology, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280